CLINICAL TRIAL: NCT02917330
Title: Stretching and Strength Training for Children With Cerebral Palsy -an Intervention Study
Brief Title: Stretching and Strength Training for Improved Gait Function in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Merete Aarsland Fosdahl, Physioteraphist, MHSc, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 519681, 2014/1766-1
Record Dates: First submitted 2016-05-11; First posted 2016-09-28 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Cerebral Palsy, Spastic, Diplegic
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strength and stretching intervention (Experimental): Treatment as usual + a strength and stretching intervention together with a physiotherapist
  Interventions: Other: Stretching and progressive strength training
- Control group (No Intervention): Treatment as usual

INTERVENTIONS:
Other: Stretching and progressive strength training — Intervention implemented by local physiotherapist.16 weeks, three treatment sessions each week. Minimum pause between two treatment sessions is one day. Week 1 and 2: To assure the correct dosage in each exercise and a satisfactory education of the session done at home, all three sessions will be implemented with the physiotherapist the first two weeks. From week 3: Two treatment/training sessions with the physiotherapist and one shorter training session at home.
  Arms: Strength and stretching intervention

SUMMARY:
The purpose of this randomized and controlled intervention study is to explore the effect of a physiotherapy intervention targeting contract and spastic hamstring muscles in children having bilateral spastic cerebral palsy (CP), GMFCS I-III: A stretching routine targeting hamstrings (and psoas if short), and a progressive strengthening program on the muscles extending then lower extremities (quadriceps, gluteus maximus and triceps surae)

Study hypothesis: Stretching of hamstrings and strength training of the extending muscles in the lower extremities in children with bilateral spastic cerebral palsy will increase popliteal angle, active knee extension, and gait function.

DETAILED DESCRIPTION:
The key intervention: 16 weeks with three treatment sessions each week. Minimum pause between two treatment sessions is one day. Week 1 and 2: To assure the correct dosage in each exercise and a satisfactory education of the session done at home, all three sessions will be implemented with the physiotherapist the first two weeks. From week 3: Two treatment/training sessions with the physiotherapist and one shorter training session at home.

Maintenance intervention: From week 17 to week nr 32.; One session pr. week will be performed at home, together with an assistant in school or with the physiotherapist. How this is accomplished will depend on what is feasible for the child and the parents.

The physiotherapy sessions: 2 sessions pr week. 5-10 min. warm up on a treadmill or a bike. A stretching exercise on the hamstrings (and psoas if shortened; ≤ 5º hip extension) and 3 strength exercises targeting the muscles extending the hip, knee and ankle.

The intervention is expected to last 30 min. and it is an extra session on top of the usual physiotherapy intervention given the child.

Home session: One session pr. week, lasting 10-15 min. No need of warm up. The session is contending one stretching exercise on hamstrings and one strength exercise. The exercises will be modified individually so the children are able to do them at home.

Exercise registration: The physiotherapist will be asked to register the sessions performed each week. The reason why a session is not performed should be registered (a scheme is attached).

The stretching (exercise schema p.3): Two stretching exercises will be performed on hamstrings, and if the psoas muscle is short (≤ 5º hip extension) there should also be a stretch performed on psoas. The stretching shall not be painful for the child.

The strength training exercises (exercises schema p.4 and 5): The strength training will be performed following the principles of "Progressive Resistance Exercise" (PRE) and the recommendations from The National Strength and Conditioning Association (NSCA) concerning strength training for children12. The recommended weight resistance for children who are familiar with strength training are 60-80% of 1RM (Repetition Maximum = maximum weight when lifting one repetition), 2- 3 sets and 8-12 repetitions, 2 -3 times per week. Verscuhen and collegues13 recommendations concerning a strength training protocol for children with CP are taken into account: not only multi -joint exercises, but also singe - joint exercises, extended rest between exercises (min 2-3 minute), minimum 12 weeks of intervention and the children should be over 7 years of age. The standing exercises shall be performed with a back pack (everyone in the intervention group will get one) which is possible to load with weights/bottles of water.

Customization of weight resistance

Children having CP are likely to be diverse and according to physical conditions and because of that 1 Repetition Maximum (1RM) will most likely be to difficult to perform. For estimation of the optimal and individualized resistance throughout the period of intervention a modified test shall be performed.

The test will be performed after the child have understood and completed the exercises correct, during the first two weeks. Until that the physiotherapist will do a mapping of the child's strength skills in order to recognize the wright amount of weight for the child for 12 repetitions and 2 series. As of week 3 there are 3 series per exercises. Recommendations from the study done by Sholtes et all14 are used for guiding of optimal weight dosage. In this study they found that for 8 RM in a sit- to stand exercise, for those having CP GMFCS I-III the weight should be 35%, 30% and 25% respectively of body weight.

Performance of the RM test: Starting out with 3 repetitions without any resistance throughout the range of moment. Every repetition shall be performed as correct and controlled as passible throughout the range of moment and the speed is 2-3 sec. per extension/flexion movement. If one repetition is carried out incorrectly with respect to speed and movement quality it shall not be counted.

The RM test shall be conducted the first time in the end of the second week (12 RM x 3 series), then next time in week 5. (10 RM x 3 series), week 8. (8 RM x 3 series), and finally in week 14. (8 RM x 3 series). When the child can do more than 12, 10 or 8 repetitions respectively, there shall be added more weight. The weight changes shall be registered in a registration form.

RM test shall be performed in exercise nr 1),2) and 3). Exercise nr 4) is mostly an awareness exercise where the focus is on quality and the ability to activate m.vastus medialis by doing a max extension in the knee in a prone position.

ELIGIBILITY:
Inclusion Criteria:

* Spastic bilateral cerebral palsy GMFCS I-III (ability to walk without aid for 10 m)
* Popliteal angle ≥ 35°

Exclusion Criteria:

* No surgical lengthening on hamstrings or bilateral triceps surae
* No surgical intervention on the lower extremities one year prior to inclusion
* No surgical intervention on the lower extremities one year prior to inclusion
* Surgical operations which is planned for the upcoming year
* No botulinum injections in hamstrings or other muscles in the lower extremities the last 6 month prior to inclusion.
* External rotation in the hips ≤ 5°
* < 90° passive ankle dorsal flexion in the ankles on a extended knee
* Reduced ability to cooperate or receive instructions

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in Hamstrings length/popliteal angle (R1 in MTS) | Measured at baseline, after 16 weeks and 32 weeks
  The tests are conducted with the child lying supine on a bench in a silent examination room and the measurements are done using a plastic goniometer, commonly used for joint and muscle measurements in the clinic.
  Two testers are doing the tests and they are a test team. If there is a contracture in the hip a pillow is placed under the knee to keep the lumbar spine straight. One tester is performing the stretch on hamstrings and the other tester is reading of the degrees on the goniometer. The pivot point for the flexion/extension axis in the knee is over the lateral condyle of femur. The aiming point for the longitudinal axis in femur is trochanter major and the aiming point for the longitudinal axis in tibia is the medial malleolus. The stationary arm on the goniometer is placed over femurs longitudinal axis and the moving arm is placed along with tibias longitudinal axis.The test is done three times and an average is calculated.

SECONDARY OUTCOMES:
Change in Active popliteal angle | Measured at baseline, after 16 weeks and 32 weeks
  This measures quadriceps ability to extend the knee into the last range of motion. It is performed in the same position as the two tests above. The child is told to stretch out the leg as much as he or she is able to (hip is hold in 90 deg by the tester). The other tester is holding the goniometer as described above and is registering the range of motion. The test is done three times and an average is calculated.
Change in Hamstrings catch (R2 modified Tardieu Scale (MTS)) | Measured at baseline, after 16 weeks and 32 weeks
  The tester is holding the actual leg, flexing the hip to 90 deg. The knee is extended and flexed slowly for two repetitions to make the child as calm and relaxed as possible, and the knee is extended fast. The quick and fast stop (catch) is measured and registered by the other tester. This test is extensively used for registration of spasticity in children with CP 18. The catch measure is only performed ones as it may change with several provocations.
Changes in Three dimensional gait analysis (3DGA) | Measured at baseline, after 16 weeks and 32 weeks
  Two skilled testers are responsible for the testing. Reflecting markers are placed on the skin according to Hellen Hays full body plug-in model. One tester is placing the markers, the other is checking and it is complete when both agree on the placement. The children are instructed to walk in a self-selected gait speed across a 10 m pathway in the lab. With infra-red light, six cameras on the wall are registrating the reflex markers attached to the children's body. The child is asked to walk back and forth between to cones placed on the floor until 5 good gait cycles is registered, meaning that the child hits two force plates in the floor by left and right foot.
Change in Cybex 6000, Strength test | Measured at baseline, after 16 weeks and 32 weeks
Changes in Pediatric quality of life questionaire 4.0 (PedsQL) | Measured at baseline, after 16 weeks and 32 weeks
  It is a self-reported Quality Of Life questionaire containing 23 questions, in 4 categories: Physical functioning, emotional functioning, social functioning and school functioning. The different themes gives a sum score between 0-100. Scale scores are computed as the sum of the items divided by the number of items answered. In addition to the four subscales, two summary scores can be computed: Physical Health Summary score (8 items) Psychosocial Health Summary score (15 items)

CONTACTS AND LOCATIONS:
Overall Officials: Inger Holm, Professor, Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No